CLINICAL TRIAL: NCT04979702
Title: Mobile Health Biometrics to Enhance Exercise and Physical Activity Adherence
Brief Title: mHealth Biometrics for Sedentary People (MotivateLJMU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Matthew Cocks, Lecturer in Muscle Biochemistry, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MotivateLJMU
Record Dates: First submitted 2021-07-16; First posted 2021-07-28 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Control (Active Comparator): Patients will have access to our online exercise resources throughout the 12-week intervention.
  Interventions: Behavioral: Active Control
- Experimental: mHealth technology assisted exercise counselling (mHealth) (Experimental): Participants will complete a 12 week mHealth technology assisted exercise counselling intervention. Participants will co-develop a 3-month structured exercise and PA programme, with support from an exercise specialist. All participants will have 4 exercise consultations with their exercise specialist. The intervention will be supported by 3 mHealth elements; 1) a wrist worn fitness watch, 2) a smartphone app for patients, and 3) a coaching website for the exercise specialist. The 3 elements will be synced, allowing data to be transferred between platforms.
  Interventions: Behavioral: mHealth technology assisted exercise counselling

INTERVENTIONS:
Behavioral: Active Control — Participants will complete a 3-month exercise and physical activity intervention supported by online recourses
  Arms: Active Control
Behavioral: mHealth technology assisted exercise counselling — Participants will complete a 3-month exercise and physical activity intervention supported by online recourses, exercise counselling sessions and mHealth technology
  Arms: Experimental: mHealth technology assisted exercise counselling (mHealth)

SUMMARY:
The investigators aim to undertake a feasibility randomised controlled trial (RCT) to investigate whether mHealth technology, allowing biometric informed feedback and coaching on exercise and PA, can be effective in previously sedentary individuals. The overall objective is to have an evidence-based exercise and PA intervention ready to evaluate in a future RCT.

DETAILED DESCRIPTION:
Participants will be recruited from Liverpool John Moores University, and other local office-based businesses. Participants will be randomised to either online exercise resources only (n=50) or exercise counselling + mHealth (n=50).This is a pilot parallel group, randomised controlled trial whereby consenting participants will complete baseline testing (T1) before starting a 12-week exercise intervention supported by online resources only (online resources intervention) or online resources and a programme of exercise counselling enhanced with mobile health (mHealth) technology (mHealth intervention). Participants will repeat baseline assessments (i) 6-weeks into the intervention (T2) and, (ii) immediately post-intervention (T3). Testing at baseline and following the 12-week intervention will include changes in physical activity, blood pressure, body composition and glycaemia control (n=20).

Both groups will have access to online resources throughout the 12-week programme. The intervention group will be provided with exercise counselling and to support this they will also be provide with a wristwatch that can monitor everyday activity and their heart rate, a smartphone app and access to a website. The intervention group will also participate in 4 consultations with an exercise specialist to plan their exercise programme and be updated on their progress towards physical activity targets. Weekly text message updates will also provide feedback to the intervention group with participants able to respond to these updates.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-75
* No known cardiovascular or metabolic disorder (e.g. heart failure, diabetes, previous myocardial infarction etc.)
* Able to exercise safely as deemed by completion of the PAR-Q+.
* Not currently meeting the recommended exercise guidelines (150 minutes moderate or 75 minutes of vigorous intensity physical activity per week), as assessed during screening questions related to the participants previous activity levels.

Exclusion Criteria:

* Aged <18 or >75
* Pregnancy or planning to become pregnant in the next 3 months
* <6 months postpartum or stopped breastfeeding <1 month before recruitment
* Not owning a smartphone with a data plan or access to WiFi

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Device derived adherence to structured exercise | Through study completion, an average 12 weeks
  Number of exercise sessions per week
Device derived duration to structured exercise | Through study completion, an average 12 weeks
  minutes of exercise completed per session
Device derived intensity of structured exercise | Through study completion, an average 12 weeks
  intensity of exercise sessions performed (% of HR max)
Change in Device derived physical activity (GENEActiv) | Baseline, Mid intervention (Week 6-7), the final 2 weeks of intervention period (weeks 10-12).
  minutes of Moderate and Vigorous physical activity
Change in Survey reported exercise behaviour (Godin Leisure Time Exercise Questionnaire (GLTEQ)) | Baseline, 4, 6, 8 12 weeks
  Bouts of mild, moderate and strenuous exercise lasting ≥30 minutes

SECONDARY OUTCOMES:
Height | Baseline, 6-weeks and immediately following intervention (12 weeks)
  Height (m)
Weight | Baseline, 6-weeks and immediately following intervention (12 weeks)
  Weight (kg)
Waist Circumference | Baseline, 6-weeks and immediately following intervention (12 weeks)
  Waist Circumference (cm)
Concentration of Hba1c | Baseline and immediately following intervention (12 weeks)
  Hba1c
Blood Lipid concentrations | Baseline and immediately following intervention (12 weeks)
  Total cholesterol, HDL/LDL, Triglycerides
Glycaemic control | Baseline and immediately following intervention (12 weeks)
  Flash glucose monitoring
Patient qualitative survey on intervention acceptability | Immediately following intervention (12 weeks)
  Study specific questionnaire (qualitative data)
Patient qualitative survey on testing acceptability | 7 Days following baseline testing
  Study specific questionnaire (qualitative data)
Exercise motivation | Baseline, Mid (week 6) and post (week 12)
  Behavioural regulation in exercise questionnaire-2 (BREQ-2). Max score 76, min score 0, high score is better
12-Item Short Form Survey | Baseline, Mid (week 6) and post (week 12)
  SF-12 Questionnaire (max 44 min 8, high score mean better outcome)
Patient Interview to access intervention acceptability | Within 2 weeks of the end of the intervention
  Patient interview
Patient Interview to access testing acceptability | Within 2 weeks of the baseline testing
  Patient interview

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share